CLINICAL TRIAL: NCT07183059
Title: Exploring Overlap Between Primary Cardiac Arrhythmias and Non-dystrophic Myotonia: a Single Center Prospective Study.
Brief Title: A Single Center Prospective Study in an Estimated 570 Patients Who Underwent Genetic Screening at UZ Brussel in the Context of a Primary Cardiac Arrhythmia. Patients Showing a Variant Class 3,4 or 5 in SCN4A or CLCN1 Will Undergo a Clinical and Electrophysiological Review After IC.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 25255_NDM-PCA studie
Record Dates: First submitted 2025-09-04; First posted 2025-09-19 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-08

CONDITIONS: Non Dystrophic Myotonia; Arrythmia, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Electromyography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exploring overlap between primary cardiac arrhythmi-as and non-dystrophic myotonia: a single center (Experimental): Patients with PCA carrying a variant class 3,4 or 5 in the SCN4A gene or a variant class 3, 4 or 5 in the CLCN1 gene will be invited by the department of Medical Genetics where they already have had a consultation, to the Neurology department for one visit on one day for the following as-sessments:
  * Interview to assess the presence, onset and duration of myotonia or episodic weakness. Assessment of medical history, family history and medical treatment.
  * Clinical neurological assessment for clinical myotonia.
  * Electromyography (EMG) to detect the presence of myotonic discharges and using the Streib and Sun score for quantification(34).
  * Short exercise test in case of myotonic discharges on nEMG.
  * In case of a diagnosis of a muscular channelopathy, assessment with.a QoL scale.
  Interventions: Diagnostic Test: Electromyography

INTERVENTIONS:
Diagnostic Test: Electromyography — we will perform questionnaire, clinical neurological exam, nEMG and if applicable short exercise test on patients with variants in genes associated with mus-cular channelopathies.
  Safety Monitoring and reporting: Needle EMG is generally well-tolerated, but transient mild proce-dural pain and discomfort are widespread and the most frequent side effect that patients will ex-perience. Hematomas are infrequent and, in most cases, asymptomatic and selflimiting. Moreover, the bleeding risk is reduced by the investigator's experience, testing superficial muscles (avoiding complications like compartment syndrome), and by not conducting an EMG when patient is treated with anticoagulants. Infectious complications at the site of needle insertion are extremely infre-quent since disposable needle electrodes are used. Needle insertion is avoided in in-jured/potential infected skin and will not be performed in immune-compromised patients and endocarditis risk.

SUMMARY:
A prospective interventional single-center study will be conducted. The study includes clinically diagnosed Intramuros PCA-patients who underwent a PCA gene panel of 113 genes (see Appendix 1) in the UZ-Brussel since 2021. In a retrospective part of the study, we will assess cardiac history, cardiac family history, cardiac exams and medical treatment and genetic data and family history. The prevalence of a class 3, 4 or 5 variant in the SCN4A and CLCN1 gene in the PCA-group will be compared to controls who underwent genetic screening for different causes, in which no association with muscular channelopathies is expected, without access to their medical file. In a prospective part of the study, patients with PCA carrying a variant class 3,4 or 5 in the SCN4A gene or a variant class 3, 4 or 5 in the CLCN1 gene will be invited for a one day visit for an interview, clinical neurological assessment and EMG. The aim of this second phase is to describe the clinical presentation of patients with concomitant PCA and non-dystrophic myotonia .

DETAILED DESCRIPTION:
A prospective interventional single-center study will be conducted. The study includes clinically diagnosed Intramuros PCA-patients who underwent a PCA gene panel of 113 genes (see Appendix 1) in the UZ-Brussel since 2021.

Retrospective part:

The following retrospective data from the medical file will be analyzed:

* Informed consents signed before genetic analysis with PCA gene panel (Appendix 2).
* Assessment of cardiac history, cardiac family history, cardiac exams and medical treatment
* Assessment of genetic data and family history.

The PCA gene panel already contains the SCN4A gene since 2021. In case patients consented to scientific research or they consented to a wide genetic testing, additional genetic screening of the CLCN1 gene will be implemented. Those who did not consent previous to the PCA-gene panel analysis, will be contacted to sign a new informed consent if interested before additional screen-ing of the CLCN1 gene.

The prevalence of a class 3, 4 or 5 variant in the SCN4A and CLCN1 gene in the PCA-group will be compared to controls who underwent genetic screening for different causes, in which no associa-tion with muscular channelopathies is expected, without access to their medical file. These con-trols are the parents of patients with a congenital malformation syndrome or patients with a neu-rodevelopmental disorder. This to evaluate whether there's a higher prevalence of skeletal muscle channelopathies in patients with PCA compared to the general population.

Prospective part:

Patients with PCA carrying a variant class 3,4 or 5 in the SCN4A gene or a variant class 3, 4 or 5 in the CLCN1 gene will be invited by the department of Medical Genetics where they already have had a consultation, to the Neurology department for one visit on one day for the following as-sessments:

* Interview to assess the presence, onset and duration of myotonia or episodic weakness. Assessment of medical history, family history and medical treatment.
* Clinical neurological assessment for clinical myotonia.
* Electromyography (EMG) to detect the presence of myotonic discharges and using the Streib and Sun score for quantification(34) (see Appendix 3).
* Short exercise test in case of myotonic discharges on nEMG.
* In case of a diagnosis of a muscular channelopathy, assessment with.a QoL scale (see Ap-pendix 4).

The aim of this second phase is to describe the clinical presentation of patients with concomitant PCA and non-dystrophic myotonia . Since there is a known clinical variability between and within families with NDM, we aim to examine whether certain clinical features or severity of the disorder are linked to cardiac involvement.

Patients of the control group, who consented for scientific research and additional testing and who consented to be informed about incidental discoveries, who carry a variant class 3,4 or 5 in the SCN4A gene or a variant class 3, 4 or 5 in the CLCN1 gene, will be invited to the Neurology de-partment for a clinical evaluation outside of the study.

Patients with a variant class 3,4 or 5 in the SCN4A gene who did beforehand not consent for scien-tific research and/or for additional genetic testing are not additionally tested for variants in the CLCN1 gene but will be invited for a clinical evaluation after consent. If,, after clinical evaluation and EMG, they are diagnosed with myotonia, additional testing for a variant in the CLCN1 gene will be proposed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PCA who underwent a genetic analysis with a PCA gene panel since 2021 (since the panel involves 112 genes including SCN4A).
* Male and female gender.

Exclusion Criteria:

* Genetic analysis before 2021
* Patients without cardiac screening in UZ Brussel

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of variants of class 3,4 or 5 in the SCN4A gene and variants of class 3, 4 or 5 in het CLCN1 gene in patients presenting with PCA. | Day 1
  the prevalence of variants of class 3,4 or 5 in the SCN4A gene and variants of class 3, 4 or 5 in het CLCN1 gene in patients presenting with PCA compared to a control group
Clinical presentation of NDMs in patients presenting with PCA and class 3,4 or 5 variants in SCN4A or CLCN1 gene. | Day 1
  the clinical presentation of NDMs in patients presenting with PCA and class 3,4 or 5 variants in SCN4A or CLCN1 gene.

IPD SHARING:
Plan to Share IPD: Undecided